CLINICAL TRIAL: NCT01040858
Title: Cognitive Rehabilitation of OIF/OEF Veterans With Cognitive Disorder
Brief Title: Cognitive Rehabilitation of Operations Iraqi Freedom and Enduring Freedom (OIF/OEF) Veterans With Cognitive Disorder
Acronym: CROVCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7217-R; IRB#2277 (Other: Portland VA Medical Center)
Record Dates: First submitted 2009-12-28; First posted 2009-12-30 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Cognition Disorders
Keywords: cognitive strategy intervention; cognitive disorders
MeSH Terms: conditions — Cognition Disorders; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Strategies Training (Experimental): Participants in the experimental group will receive the Cognitive strategy intervention during the first ten weeks of their participation in the study, whereas comparison group participants will continue to receive usual care (no cognitive strategy intervention) during their participation in the study (but will be offered cognitive strategy intervention after the end of the study). Cognitive Strategies training consisted of interactive didactic presentations, in-class discussions, and activities that introduced participants to a variety of cognitive strategies and external aids.
  Interventions: Behavioral: Cognitive Strategy Training
- Placebo comparison group (Placebo Comparator): Participants in the experimental group will receive the Cognitive strategy intervention during the first ten weeks of their participation in the study, whereas comparison group participants will continue to receive usual care (no cognitive strategy intervention) during their participation in the study (but will be offered cognitive strategy intervention after the end of the study).
  Interventions: Other: Placebo comparison group

INTERVENTIONS:
Behavioral: Cognitive Strategy Training — Cognitive Strategy Training will consist of weekly 120-minute group sessions for 10 weeks.
  Arms: Cognitive Strategies Training
Other: Placebo comparison group — Participants in the experimental group will receive the Cognitive strategy intervention during the first ten weeks of their participation in the study, whereas comparison group participants will continue to receive usual care (no cognitive strategy intervention) during their participation in the study (but will be offered cognitive strategy intervention after the end of the study).
  Arms: Placebo comparison group

SUMMARY:
The number of OEF/OIF veterans seeking care and rehabilitation services within the VA Health Care System is increasing rapidly. The cognitive effects of MTBI are clinically significant and can adversely affect a veteran's ability to reintegrate into civilian life, return to duty, succeed in competitive employment, or function independently. The primary product of the proposed study would be an empirically validated, manualized, cognitive rehabilitation intervention for OIF/OIF veterans with cognitive disorders. The group treatment modality has the virtue of efficiency and a manualized treatment approach would allow wide-ranging application throughout the VHA system. As such, the proposed study is likely to have a significant effect on the quality and effectiveness of rehabilitative services being offered to our returning soldiers with combat-related MTBI and cognitive impairment.

DETAILED DESCRIPTION:
As a result of the current military operations in Afghanistan (Operation Enduring Freedom; OEF) and Iraq (Operation Iraqi Freedom; OIF), the Department of Veterans Affairs (VA) is providing health care for increasing numbers of veterans who have experienced mild traumatic brain injury (MTBI) or concussion, many of whom complain of cognitive impairment. MTBI is the most common combat-related injury and can occur with or without direct impact, obvious external injuries, or loss of consciousness. Currently, cognitive rehabilitation for MTBI typically includes training in compensatory strategies that help patients develop internal strategies (e.g., visual imagery) and utilize external aides (e.g., memory notebooks, calendars/organizers, timers) to compensate for cognitive deficits. Initial data from our unfunded cognitive rehabilitation pilot study are encouraging and indicate post-treatment improvement on multiple outcome measures. However, to date, no published studies have evaluated the efficacy of specific cognitive rehabilitation interventions with OEF/OIF veterans who have experienced combat-related MTBI. The primary objective of this study, therefore, is to evaluate the efficacy of a manualized, 10-week, Compensatory Strategy Training (CST) intervention for OEF/OIF veterans with cognitive disorder resulting from the aftereffects of combat-related mild traumatic brain injury. The specific goals are: 1) to determine the efficacy of cognitive rehabilitation group treatment; and 2) to determine the treatment factors and patient characteristics that are associated with improved functional outcomes. The overall goal is to develop an evidence-based, manualized, group treatment that can be readily implemented in VHA treatment settings. The study design makes use of the convergent availability of resources available at the four participating VAs in Portland Oregon, Puget Sound Washington, San Diego California, and Boise Idaho. The study will recruit a total of 280 OEF/OIF veterans enrolled for medical services at these VAs. In a randomized controlled trial, we will compare two groups: eligible participants will be randomly assigned to either the Cognitive Strategy Training (CST) group or Usual Care (UC) group. Participants in the CST group will receive the CST intervention during their participation in the study, which will consist of weekly 120-minute group sessions for 10 weeks as guided by the CST Treatment Manual. UC participants will continue to receive usual care (i.e., their regular medical, psychiatric, and psychotherapeutic care; no CST intervention) during their participation, but will be offered CST after the end of the study. Both groups will undergo assessments at baseline, 5 weeks (midway through CST),10 weeks (immediately following the end of CST), and 15 weeks (5 weeks after CST is completed). These assessments will include a brief cognitive assessment battery and a battery of questionnaires and paper-pencil tests designed to assess current psychological and cognitive symptom severity, utility of compensatory strategies, self-efficacy, adaptive functioning, ability to reliably manage personal affairs, substance use, quality of life, and treatment satisfaction ratings. During their study participation, all participants will continue to receive their regular medical, psychiatric, and psychotherapeutic care.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF veterans enrolled at a participating VA who are able to provide informed consent; and
* As part of standard VA clinical care, have screened positive for MTBI and complain of cognitive impairment.

Exclusion Criteria:

* Current substance use disorder with less than 30 days abstinence;
* History of a primary psychotic disorder; and
* Auditory or visual impairments that would prevent ability to participate in the cognitive rehabilitation group or benefit from compensatory strategies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Storzbach, PhD, Principal Investigator — VA Medical Center, Portland
Locations (4):
- United States (4):
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - VA Medical Center, Boise, Boise, Idaho
  - VA Medical Center, Portland, Portland, Oregon
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington

REFERENCES:
- [Derived] Pagulayan KF, O'Neil M, Williams RM, Turner AP, Golshan S, Roost MS, Laman-Maharg B, Huckans M, Storzbach D, Twamley EW. Mental Health Does Not Moderate Compensatory Cognitive Training Efficacy for Veterans With a History of Mild Traumatic Brain Injury. Arch Phys Med Rehabil. 2017 Sep;98(9):1893-1896.e2. doi: 10.1016/j.apmr.2017.04.009. Epub 2017 May 5. PMID 28483653

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Strategies Training: Participants in the experimental group received the Cognitive Strategies intervention during their participation in the study. Cognitive Strategies Training consisted of weekly 120-minute group sessions for 10 weeks.
- Placebo Comparison Group: Placebo comparison group continued to receive usual care and did not receive Cognitive Strategies training duirng their participation in the study. They were, however, offered to receive the training at the end of their participation in the study.
Period: Overall Study
Arm/Group | Cognitive Strategies Training | Placebo Comparison Group
Started | 59 | 69
Completed | 50 | 69
Not Completed | 9 | 0

BASELINE CHARACTERISTICS:
Population: Of the 128 subjects who consented to participate in the study, 9 participants who were randomized to the Cognitive Strategies Training, did not complete the training due to schedule conflict, etc. Thus, their data was not included in the final analysis.
Groups:
- Cognitive Strategies Group: Participants in the experimental group received the Cognitive Strategies intervention during their participation in the study. Cognitive Strategies Training consisted of weekly 120-minute group sessions for 10 weeks.
- Total: Total of all reporting groups
Arm/Group | Cognitive Strategies Group | Placebo Comparison Group | Total
Number analyzed (Participants) | 50 | 69 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (7) | 35.4 (8) | 34.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 47 | 66 | 113
The Neurobehavioral Symptom Inventory [Mean (Standard Deviation); unit: units on a scale] — A post-concussive symptom measure. The total score on the measure is the sum of severity ratings for 22 symptoms on a scale from 0 (none) to 4 (very severe). NSI total score ranges from 0 to 88.
  units on a scale | 45.04 (16.32) | 44.8 (14.5) | 44.90 (14.01)
Prospective-Retrospective Memory Questionnaire [Mean (Standard Deviation); unit: units on a scale] — A 16-item self-report severity measure of prospective and retrospective memory problems relevant to everyday life. The measure reports the sum of severity ratings on a scale from 1 (never) to 5 (very often). The PRMQ total score ranges from 16 to 80.
  units on a scale | 57.2 (8) | 55.4 (10) | 56.1 (9.5)
Multiple Sclerosis Neuropsychological Screening Questionnaire-Patient Version [Mean (Standard Deviation); unit: units on a scale] — A self-report measure of severity of attention and organizational problems. It measures the sum of severity ratings on a scale from 0 (never) to 4 (very often). The total score ranges from 0 to 64.
  units on a scale | 37.8 (9) | 37.0 (10) | 37.3 (9.7)
Memory Compensation Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The MCQ is a 44-item self-report questionnaire that rates the extent to which patients use various strategies to improve memory performance relevant to daily living. The MCQ measures the sum of memory strategies used on a scale from 0 (never) to 4 (always). The total score ranges from 0 to 176.
  units on a scale | 119.8 (24) | 118.5 (7) | 119.03 (24.7)
The Wide Range Achievement Test-IV [Mean (Standard Deviation); unit: units on a scale] — Reading subtest that provides an estimate of baseline cognitive ability. This assessment was administered only at baseline, and was not repeated. The total score ranges from 55 (lower cognitive ability) to 145 (higher cognitive ability).
  units on a scale | 97.02 (8.75) | 99.70 (8.3) | 98.56 (8.6)
Hopkins Verbal Memory Test-Revised [Mean (Standard Deviation); unit: units on a scale] — Verbal list learning and delayed recall. Total recall T-score was used for the analyses. Total recall T-score ranges from 13 (severely impaired) to 86 (very superior).
  units on a scale | 41.6 (11.2) | 40.48 (12.2) | 40.95 (11.7)
Wechsler Adult Intelligence Scale-Digit Span [Mean (Standard Deviation); unit: units on a scale] — A measure of attention and working memory. Total score was used, and it ranges from 0 to 48, with higher scores indicating greater attentional capacity.
  units on a scale | 25.76 (5.42) | 27.10 (6.41) | 26.53 (6.0)
Delis-Kaplan Executive Function System, Trails Subtest [Mean (Standard Deviation); unit: units on a scale] — A visual-motor task used to measure flexibility in thinking (executive function) and processing speed. Scaled score for Condition 4 was used, and possible scores ranges from 0 to 20 with higher scores indicating better outcome.
  units on a scale | 9.3 (3) | 9.84 (2) | 9.31 (3)
Delis-Kaplan Executive Function System, Letter Fluency Subtest [Mean (Standard Deviation); unit: units on a scale] — A measure of verbal fluency, generativity, and processing speed. A scaled score of Letter Fluency portion of the test was used. The scores ranged from 0 to 20 with higher scores indicating better outcomes.
  units on a scale | 9.78 (3.3) | 10.18 (3.7) | 10.01 (3.5)
PTSD Checklist-Military Version [Mean (Standard Deviation); unit: units on a scale] — A PTSD symptom severity measures based on DSM-IV diagnostic criteria. It measures the sum of severit ratings for 17 symptoms on a scale from 1 (not at all) to 5 (extremely). PCL-M total score ranges from 17 to 85.
  units on a scale | 57.50 (14.5) | 58.94 (14.5) | 58.31 (14.4)
Beck Depression Inventory, Second Edition [Mean (Standard Deviation); unit: units on a scale] — A depression symptom severity measures based on DSM-IV diagnostic criteria. It measures the sum of severity ratings for 21 symptoms on a scale from 0 (none) to 3 (severe). BDI total score ranges from 0 to 63.
  units on a scale | 24.9 (12.2) | 25.3 (12.6) | 25.11 (12.34)
Severity of Dependence Scale [Mean (Standard Deviation); unit: units on a scale] — A brief substance dependence measure. It measures the sum of severity ratings for 5 symptoms on a scale from 0 (never) to 3 (always). The total score ranges from 0 15.
  units on a scale | 1.04 (2.3) | 0.46 (1.2) | 0.70 (1.78)
Satisfaction with Life Scale [Mean (Standard Deviation); unit: units on a scale] — A brief measure of global life satisfaction. It measures the sum of satisfaction ratings for 5 items on a scale from 1 (strongly disagree) to 7 (strongly agree). The total score ranges from 5 to 35 with higher scores indicating greater satifaction.
  units on a scale | 16.30 (7.5) | 16.73 (7.1) | 16.6 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Multiple Sclerosis Neuropsychological Screening Questionnaire-Patient Version
Description: A self-report measure of severity of attention and organizational problems. It measures the sum of severity ratings on a scale from 0 (never) to 4 (very often). The total score ranges from 0 to 64.
Time Frame: Week 10
Population: The number of participants who completed this measure at Week 10 was lower than baseline due to missing data, or incomplete data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Strategies Training | Placebo Comparison Group
Number analyzed (Participants) | 36 | 51
units on a scale | 33.58 (9.52) | 36.35 (10.23)

2. Secondary Outcome: Prospective-Retrospective Memory Questionnaire (PRMQ; Crawford, Henry, Ward, &
Description: A 16-item self-report severity measure of prospective and retrospective memory problems relevant to everyday life. The measure reports the sum of severity ratings on a scale from 1 (never) to 5 (very often). The PRMQ total score ranges from 16 to 80.
Time Frame: Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Strategies Training | Placebo Comparison Group
Number analyzed (Participants) | 36 | 51
units on a scale | 49.56 (10) | 55.20 (12)

3. Secondary Outcome: The Neurobehavioral Symptom Inventory
Description: A post-concussive symptom measure. The total score on the measure is the sum of severity ratings for 22 symptoms on a scale from 0 (none) to 4 (very severe). NSI total score ranges from 0 to 88.
Time Frame: Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo comparison group continued to receive usual care and did not receive Cognitive Strategies training duirng their participation in the study. They were, however, offered to receive the training at the end of their participation in the study.
Arm/Group | Cognitive Strategies Training | Placebo
Number analyzed (Participants) | 36 | 52
units on a scale | 40.89 (17.7) | 43.52 (17.69)

4. Secondary Outcome: Memory Compensation Questionnaire
Description: The MCQ is a 44-item self-report questionnaire that rates the extent to which patients use various strategies to improve memory performance relevant to daily living. The MCQ measures the sum of memory strategies used on a scale from 0 (never) to 4 (always). The total score ranges from 0 to 176.
Time Frame: Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Participants in the experimental group received the Cognitive Strategies intervention during their participation in the study. Cognitive Strategies Training consisted of weekly 120-minute group sessions for 10 weeks.
- Arm 2: Placebo comparison group continued to receive usual care and did not receive Cognitive Strategies training duirng their participation in the study. They were, however, offered to receive the training at the end of their participation in the study.
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 36 | 52
units on a scale | 123.08 (26.2) | 119.52 (28.33)

5. Secondary Outcome: Hopkins Verbal Memory Test-Revised
Description: Verbal list learning and delayed recall. Total recall T-score was used for the analyses. Total recall T-score ranges from 13 (severely impaired) to 86 (very superior).
Time Frame: Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Strategies Training | Placebo
Number analyzed (Participants) | 36 | 51
units on a scale | 50.50 (12.97) | 44.75 (12.2)

6. Secondary Outcome: Wechsler Adult Intelligence Scale-3rd Edition, Digit Span Subtest
Description: A measure of attention and working memory. Total score was used, and it ranges from 0 to 48, with higher scores indicating greater attentional capacity.
Time Frame: Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Strategies Training | Placebo
Number analyzed (Participants) | 36 | 52
units on a scale | 28.39 (5.76) | 28.58 (5.79)

7. Secondary Outcome: Delis-Kaplan Executive Function System, Trails Subtest
Description: A visual-motor task used to measure flexibility in thinking (executive function) and processing speed. Scaled score for Condition 4 was used, and possible scores ranges from 0 to 20 with higher scores indicating better outcome.
Time Frame: Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Strategies Training | Placebo
Number analyzed (Participants) | 36 | 52
units on a scale | 9.89 (2.9) | 10.38 (2.24)

8. Secondary Outcome: Delis-Kaplan Executive Function System, Verbal Fluency Subtest
Description: A measure of verbal fluency, generativity, and processing speed. A scaled score of Letter Fluency portion of the test was used. The scores ranged from 0 to 20 with higher scores indicating better outcomes.
Time Frame: Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Strategies Training | Placebo
Number analyzed (Participants) | 36 | 52
units on a scale | 11.31 (2.72) | 10.63 (3.10)

9. Secondary Outcome: PTSD Checklist-Military Version
Description: A PTSD symptom severity measures based on DSM-IV diagnostic criteria. It measures the sum of severit ratings for 17 symptoms on a scale from 1 (not at all) to 5 (extremely). PCL-M total score ranges from 17 to 85.
Time Frame: Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Strategies Training | Placebo
Number analyzed (Participants) | 36 | 50
units on a scale | 53.22 (16.42) | 57.18 (17.0)

10. Secondary Outcome: Beck Depression Inventory, Second Edition
Description: A depression symptom severity measures based on DSM-IV diagnostic criteria. It measures the sum of severity ratings for 21 symptoms on a scale from 0 (none) to 3 (severe). BDI total score ranges from 0 to 63.
Time Frame: Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Strategies Training | Placebo
Number analyzed (Participants) | 36 | 52
units on a scale | 20.53 (14) | 23.75 (14.79)

11. Secondary Outcome: Severity of Dependence Scale
Description: A brief substance dependence measure. It measures the sum of severity ratings for 5 symptoms on a scale from 0 (never) to 3 (always). The total score ranges from 0 15.
Time Frame: Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Strategies Training | Placebo
Number analyzed (Participants) | 36 | 51
units on a scale | 0.67 (2.01) | 0.73 (2.1)

12. Secondary Outcome: Satisfaction With Life Scale
Description: A brief measure of global life satisfaction. It measures the sum of satisfaction ratings for 5 items on a scale from 1 (strongly disagree) to 7 (strongly agree). The total score ranges from 5 to 35 with higher scores indicating greater satifaction.
Time Frame: Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Strategies Training | Placebo
Number analyzed (Participants) | 36 | 52
units on a scale | 17.44 (8.5) | 17.69 (7.8)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/69
Other Adverse Events (participants affected / at risk) | 0/50 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No